CLINICAL TRIAL: NCT04055337
Title: Flap Sliding Technique for Managing Flap Striae Following Laser in Situ Keratomileusis
Brief Title: Flap Sliding to Treat Post-LASIK Striae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate Professor of Ophthalmology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17300292
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: LASIK Complication Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flap Sliding (Experimental): noninvasive "flap sliding" technique for managing flap striae following laser in situ keratomileusis (LASIK).
  Interventions: Procedure: Flap sliding

INTERVENTIONS:
Procedure: Flap sliding — All subjects underwent the "flap sliding" technique, which was performed at the Alforsan Eye Centre in Assiut, Egypt. Prior to surgery, all subjects underwent corneal imaging with anterior segment optical coherence tomography to confirm the presence of striae. All surgical procedures were performed by the same surgeon 1 or 2 days following LASIK.
  Subjects were administered a topical anesthetic. Striae location and orientation were then determined after drying the corneal surface with a cellulose sponge. The sponge was used to push the LASIK flap over the stromal bed in a direction that was perpendicular to the striae. The flap was pushed from the proximal side of the striae toward the flap edge. The ultimate goal was to move striae and put the flap into its proper place. Following surgery, OCT imaging was repeated.

SUMMARY:
This study assessed the efficacy and safety of a simple, noninvasive "flap sliding" technique for managing flap striae following laser in situ keratomileusis (LASIK). Included eyes underwent flap sliding 1-2 days after surgery, which involved using a cellulose sponge to gently slide the flap perpendicular to the striae. The flap was not lifted during the procedure. Thirteen of 14 eyes were successfully managed with flap sliding. Uncorrected distance visual acuity (DVA) improved in all patients 1 day after flap sliding, with 11 eyes having a corrected DVA of 20/25 or better. Complications following flap sliding occurred in 2 eyes. We believe that our study makes a significant contribution to the literature because it demonstrates a simple, noninvasive technique for managing flap striae that develop during early post-LASIK epithelial healing.

ELIGIBILITY:
Inclusion Criteria:

Significant flap striae in the visual zone within 2 days following microkeratome LASIK.

Exclusion Criteria:

* striae 2 days after surgery
* visually insignificant striae

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
UDVA | 1 day
  Uncorrected distance visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Alforsan eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelazeem K, Nassr MA, Abdelmotaal H, Wasfi E, El-Sebaity DM. Flap Sliding Technique for Managing Flap Striae following Laser In Situ Keratomileusis. J Ophthalmol. 2020 Feb 24;2020:5614327. doi: 10.1155/2020/5614327. eCollection 2020. PMID 32185074